CLINICAL TRIAL: NCT02456142
Title: EFFECT OF CAUDAL BUPIVACAINE VERSUS INTRAVENOUS MORPHINE ON TIME TO FIRST ANALGESIC REQUIREMENT IN PEDIATRIC SURGICAL PATIENTS; A RANDOMISED CONTROLLED TRIAL.
Brief Title: CAUDAL BUPIVACAINE VERSUS INTRAVENOUS MORPHINE ON TIME TO FIRST ANALGESIC REQUIREMENT
Acronym: CaBuMorph
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Makerere University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206005358
Record Dates: First submitted 2015-05-25; First posted 2015-05-28 (Estimated); Last update posted 2016-04-11 (Estimated); Status verified 2015-05

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- caudal bupivacaine (Experimental): 1ml/kg of 0.125% caudal bupivacaine given over 2 minutes will be given at the end of surgery
  Interventions: Drug: caudal bupivacaine
- intravenous morphine (Active Comparator): 0.05mg/kg intravenous morphine given over 5 minutes
  Interventions: Drug: intravenous morphine

INTERVENTIONS:
Drug: caudal bupivacaine
  Other Names: BUPICAN Heavy
  Arms: caudal bupivacaine
Drug: intravenous morphine
  Arms: intravenous morphine

SUMMARY:
Pain is a subjective sensation which in children can only be experienced and most times not expressed. Pain management in children thus falls short of their adult counterparts. Acute pain of surgery causes significant suffering and stress. In children, pain management has lagged behind because of the belief that children's pain receptors are less well developed than their adult counterparts. However this has been proven to be false as development of pain receptors has been shown by 26th week of gestation. Caudal analgesia with plain bupivacaine has been used for effective post operative analgesia. Resources sometimes limit acquisition of additives to bupivacaine to be delivered into the intrathecal space.

The fear of pharmacological adverse effects of opioids has restricted their use especially among the anesthesia officers who deliver the bulk of anesthesia services in Uganda and this has led to poor pain management in pediatric populations Mulago national referral hospital is a resource limited centre with regards to human resource, equipment and drugs. This is mainly due to lack of sufficient funds and large volume of patients with the nursing staff being overwhelmed by the patient capacity. Drug administration is often not done on time and continuous assessment of pain scores in children is not adequate resulting in poor post operative pain management. Pain control thus will depend on analgesia provided at the time of operation creating a need for prolonged pain control measures.

Studies done have compared intravenous morphine administration versus caudal analgesia and are mostly focused of sub umbilical surgery however none has been done in our setting. Bupivacaine and morphine are now more readily available and can be used for post operative analgesia. However studies on the timing to the next analgesic requirement have not been compared/done in Mulago national referral hospital.

DETAILED DESCRIPTION:
Patients will be wheeled into the operating theatre.

* Anaesthesia will be induced using an inhalation anaesthetic (sevoflurane) and intravenous anaesthetic using propofol or thiopental for the older children (3 years and above).
* Maintenance of anaesthesia will be done using either inhalation anaesthetic (sevoflurane)
* Intra-operative analgesia will be maintained with intravenous fentanyl given at the start of surgery and hourly for surgeries longer than one hour.
* Monitoring intra and post operatively will be done with WHO standard monitoring. (Blood pressure, heart rate, saturation, temperature, ECG, End tidal carbon dioxide).
* The intervention will be given at the end of surgery after the last stitch has been placed with patient receiving either caudal bupivacaine or intravenous morphine.
* to receive a caudal the baby will be placed in the left lateral position knees and hips flexed
* The skin over the coccyx and sacrum will be cleansed with povidone-iodine solution and alcohol.
* After palpation of the sacral cornua, a 22- or 23-gauge needle will be placed into the sacral hiatus to identify the epidural space by loss of resistance as the needle passes through the sacral ligament.
* Aspiration will be done to check for cerebrospinal fluid or blood, then a test dose is administered to rule out intravenous injection then the drug caudal bupivacaine will be injected.
* The patients' pain scores will be assessed by the research assistant in the post anaesthesia care unit after 30 minutes before being discharged to their parent wards and hourly after the intervention is given.
* monitoring of pulse rate and saturation on the ward will be done with a pulse oximeter.
* On the ward the pain scores will be assessed every hour by the research assistant and time to a pain score of 4 recorded
* The pain scores and the time to the next analgesic requirement will be recorded and continuation of analgesia given with intravenous paracetamol.

The crying, requires oxygen, increased vital signs, expression, sleeplessness (CRIES) pain tool will be used to score pain in neonates and the Face, Legs, Activity, Cry and Consolability (FLACC) pain score used in children above 2 months. Analgesic requirement will be given if child found to be in pain.

ELIGIBILITY:
Inclusion Criteria:

- All American Society of Anesthesia (ASA )I and II patients aged less than 8years undergoing elective abdominal perineal and lower limb orthopedic surgery

Exclusion Criteria:

* Known hypersensitivity to opioids Known hypersensitivity to local anesthetics

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
time to first analgesic requirement | 24 hours
  time from intervention to pain score of 4
Post- operative pain scores of the patients using age appropriate scales. | 24 hours
  comparing the pain scores of the patients using the FLACC and the CRIES pain tools

SECONDARY OUTCOMES:
Adverse effects reactions of the intravenous morphine analgesia and caudal analgesia | 24 hours
  watch for respiratory depression,anaphylaxis

CONTACTS AND LOCATIONS:
Overall Officials: EZRA MUGISHA, MBChB, Principal Investigator — makerere university college of health sciences department of anesthesia
Locations (1):
- Mulago Hospital Complex, Kampala, Kampala, Uganda